CLINICAL TRIAL: NCT02946866
Title: A Prospective Study for the Natural History and the Risk Factors of Prospective Symptomatic Hemorrhage in Adult Patients With Cerebral Cavernous Malformation
Brief Title: CoHOrt of Cerebral CavernOus maLformATion: multicEnter Prospective Observational Study
Acronym: CHOCOOATE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); KangWon National University Hospital (Other); Jeju National University Hospital (Other); Chuncheon Sacred Heart Hospital (Other); SMG-SNU Boramae Medical Center (Other); Gyeongsang National University Hospital (Other); Soonchunhyang University Hospital (Other); Johannes Gutenberg University Mainz (Other); First Affiliated Hospital of Suzhou Medical College (Other)
Responsible Party: Principal Investigator, Jeong Eun Kim, Professor, Seoul National University Hospital
Other Study IDs: SNUH-002
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Cavernous Malformation; Intracerebral Hemorrhage
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cerebral cavernous malformation: Patients with newly diagnosed, cerebral cavernous malformation who will visit one of the study centers during the period from June 2016 to December 2017. Patients would be eligible for enrollment if they were 18 years of age or older and had at least 1 cavernous malformation. All patients who would visit a study center during the enrollment period and meet these criteria will be asked to join the study. The cohort will consists of patients who agree to participate. Target population of this study is 228 patients.

SUMMARY:
The aim of this prospective study is to reveal the natural history of symptomatic hemorrhage in adult patients with cerebral cavernous malformation with the goal of informing the treatment plan.

DETAILED DESCRIPTION:
Cerebral cavernous malformation Patients with newly diagnosed, cerebral cavernous malformation who will visit one of the study centers during the period from June 2016 to December 2017. Patients would be eligible for enrollment if they were 18 years of age or older and had at least 1 cerebral cavernous malformation. If the patient had multiple cavernous malformations, index cavernous malformation would be enrolled. Index lesion will be determined according to the criteria.

* Index lesion decision criteria I. Symptomatic II. Asymptomatic (priorities are as follows)

  1. Previous bleed
  2. Brain stem location
  3. Deep nuclei (thalamus, caudate, basal ggl, hypothalamus)
  4. Periventricular
  5. Largest

All patients who would visit a study center during the enrollment period and meet these criteria will be asked to join the study. The cohort will consists of patients who agree to participate. Target population of this study is 228 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed cerebral cavernous malformation who agreed to participate.
* 18 years old or more

Exclusion Criteria:

* Patients who underwent treatment(surgery or radiosurgery) for cavernous malformation
* Patients who are accompanied by other serious medical problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators defined the cohort population as adults( more than 18 years old) with newly diagnosed cerebral cavernous malformation who agree to participate.
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2016-06; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic hemorrhage | 5 year
  hemorrhage due to rupture of cavernous malformation

SECONDARY OUTCOMES:
Symptomatic hemorrhage | 1 year
  hemorrhage due to rupture of cavernous malformation
All hemorrhagic event including radiologic rupture + newly appeared neurologic symptom | 1 year
  hemorrhage without symptom
All hemorrhagic event including radiologic rupture | 5 year
  all hemorrhagic events

CONTACTS AND LOCATIONS:
Overall Officials: JeongEun Kim, MD. PhD., Principal Investigator — Study Principal Investigator
Locations (8):
- South Korea (8):
  - KangWon National University Hospital, Chuncheon, Gangwon-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - HUMC-Chuncheon Sacred Heart Hospital, Chuncheon, Kanwon
  - DongGuk University, Ilsan, Kyungkido
  - Jeju National University Hospital, Jeju City
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeon JS, Kim JE, Chung YS, Oh S, Ahn JH, Cho WS, Son YJ, Bang JS, Kang HS, Sohn CH, Oh CW. A risk factor analysis of prospective symptomatic haemorrhage in adult patients with cerebral cavernous malformation. J Neurol Neurosurg Psychiatry. 2014 Dec;85(12):1366-70. doi: 10.1136/jnnp-2013-306844. Epub 2014 Mar 28. PMID 24681702
- [Background] Horne MA, Flemming KD, Su IC, Stapf C, Jeon JP, Li D, Maxwell SS, White P, Christianson TJ, Agid R, Cho WS, Oh CW, Wu Z, Zhang JT, Kim JE, Ter Brugge K, Willinsky R, Brown RD Jr, Murray GD, Al-Shahi Salman R; Cerebral Cavernous Malformations Individual Patient Data Meta-analysis Collaborators. Clinical course of untreated cerebral cavernous malformations: a meta-analysis of individual patient data. Lancet Neurol. 2016 Feb;15(2):166-173. doi: 10.1016/S1474-4422(15)00303-8. Epub 2015 Dec 2. PMID 26654287
- [Background] Al-Shahi Salman R, Berg MJ, Morrison L, Awad IA; Angioma Alliance Scientific Advisory Board. Hemorrhage from cavernous malformations of the brain: definition and reporting standards. Angioma Alliance Scientific Advisory Board. Stroke. 2008 Dec;39(12):3222-30. doi: 10.1161/STROKEAHA.108.515544. Epub 2008 Oct 30. PMID 18974380
- [Background] Porter PJ, Willinsky RA, Harper W, Wallace MC. Cerebral cavernous malformations: natural history and prognosis after clinical deterioration with or without hemorrhage. J Neurosurg. 1997 Aug;87(2):190-7. doi: 10.3171/jns.1997.87.2.0190. PMID 9254081
- [Background] Flemming KD, Link MJ, Christianson TJ, Brown RD Jr. Prospective hemorrhage risk of intracerebral cavernous malformations. Neurology. 2012 Feb 28;78(9):632-6. doi: 10.1212/WNL.0b013e318248de9b. Epub 2012 Feb 1. PMID 22302553
- [Background] Schneble HM, Soumare A, Herve D, Bresson D, Guichard JP, Riant F, Tournier-Lasserve E, Tzourio C, Chabriat H, Stapf C. Antithrombotic therapy and bleeding risk in a prospective cohort study of patients with cerebral cavernous malformations. Stroke. 2012 Dec;43(12):3196-9. doi: 10.1161/STROKEAHA.112.668533. Epub 2012 Nov 13. PMID 23150651
- [Background] Al-Shahi Salman R, Hall JM, Horne MA, Moultrie F, Josephson CB, Bhattacharya JJ, Counsell CE, Murray GD, Papanastassiou V, Ritchie V, Roberts RC, Sellar RJ, Warlow CP; Scottish Audit of Intracranial Vascular Malformations (SAIVMs) collaborators. Untreated clinical course of cerebral cavernous malformations: a prospective, population-based cohort study. Lancet Neurol. 2012 Mar;11(3):217-24. doi: 10.1016/S1474-4422(12)70004-2. Epub 2012 Jan 31. PMID 22297119